CLINICAL TRIAL: NCT06616974
Title: A Phase 2, Double-blind, Randomized, Placebo-Controlled Study to Assess the Efficacy and Safety of TX000045 After 24 Weeks of Treatment in Patients With Pulmonary Hypertension Secondary to Heart Failure With Preserved Ejection Fraction (PH-HFpEF)
Brief Title: A Study of TX000045 in Patients With Pulmonary Hypertension Secondary to Heart Failure With Preserved Ejection Fraction (the APEX Study)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tectonic Therapeutic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TX000045-003
Record Dates: First submitted 2024-09-19; First posted 2024-09-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TX000045 Dose A (Experimental): Participants will receive a single dose of TX000045 Dose A subcutaneously every 2 weeks for 24 weeks from Day 1 to Day 155.
  Interventions: Drug: TX000045- Dose A
- TX000045 Dose B (Experimental): Participants will receive alternating single doses of TX000045 Dose B and placebo subcutaneously every 2 weeks for 24 weeks from Day 1 to Day 155.
  Interventions: Drug: TX000045- Dose B
- Placebo (Placebo Comparator): Participants will receive a single placebo dose SC for 24 weeks from Day 1 to Day 155
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TX000045- Dose A — The participants will receive a subcutaneous injection of Dose A of TX000045 every 2 weeks for 24 weeks.
  Arms: TX000045 Dose A
Drug: TX000045- Dose B — The participants will receive subcutaneous injection of Dose B of TX000045 every 4 weeks for 24 weeks where they will alternate between TX000045 and placebo every 2 weeks.
  Arms: TX000045 Dose B
Drug: Placebo — The participants will receive a subcutaneous injection of placebo every 2 weeks for 24 weeks.
  Arms: Placebo

SUMMARY:
TX000045-003 is a double-blind, randomized, parallel group, placebo-controlled, proof- of-concept (POC) study, evaluating 2 dose regimens of TX000045 over the course of a 24-week treatment period (the APEX study).

DETAILED DESCRIPTION:
This study will enroll approximately 180 participants and eligible patients will be randomized to one of 3 treatment arms:

* Arm 1: Treatment Group 1: Placebo delivered subcutaneously (SC) every 2 weeks (Q2W) for 24 weeks
* Arm 2: Treatment Group 2: TX000045 SC at Dose A Q2W for 24 weeks
* Arm 3: Treatment Group 3: TX000045 SC at Dose B Q2W alternating with Placebo Q2W for 24 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female of non-childbearing potential between the ages of 18 and 83 years.
2. Has a diagnosis of PH-HFpEF based on baseline echocardiogram and right heart catheterization (RHC).
3. Has NYHA functional class II- III heart failure.
4. Has 6MWT distance from 100 to 450m.
5. Chronic medication for heart failure or cardiovascular disease is at a stable dose prior to screening.
6. Is able to understand and provide documented consent for participation.

Exclusion Criteria:

1. Diagnosis of PH in World Health Organization (WHO) Group 1, WHO Group 3, WHO Group 4, or WHO Group 5.
2. Current or recent hospitalization prior to screening.
3. Recently received vasoactive drugs, pulmonary arterial hypertension-specific therapies, or a relaxin receptor agonist.
4. Initiated a new exercise program for cardiopulmonary rehabilitation or plans to initiate such a program during the study.
5. Has a body mass index <18 kg/meter square or >45 kg/ meter square.
6. Was previously administered TX000045, relaxin, or a relaxin fusion protein.
7. Historical or current evidence of a clinically significant disease or disorder such as significant lung disease, cardiovascular comorbitiies, liver disease, infectious disease, or malignancy.
8. Has any of the following clinical laboratory values during screening:

   1. Serum alanine aminotransferase or aspartate aminotransferase levels > 3 x the upper limit of normal (ULN) or total bilirubin > 3 x ULN;
   2. eGFR <30 mL/min/1.73 m2;
   3. HbA1c (glycosylated hemoglobin) >9%;
   4. Platelet count <50,000/millimeter cube;
   5. Hemoglobin <10.0g/dL;
9. History of hypersensitivity or reactions to drugs with a similar chemical structure or class to TX000045.
10. Is pregnant or breastfeeding.
11. Has a history of cancer within 5 years of screening other than basal cell carcinoma, cervical carcinoma, or squamous cell carcinomas of the skin.
12. Has a history of drug or alcohol abuse.
13. Was recently dosed in any clinical research study.

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Pulmonary Vascular Resistance (PVR) in participants with a combined pre- and post-capillary pulmonary hypertension (CpcPH). | Baseline up to Week 24 post first dose
  Measured by right heart catheterization (RHC) between those who received TX000045 and those with placebo.
Assess safety of TX000045 by the incidence of adverse events, adverse events of special interest and SAEs. | Baseline up to Week 30 post first dose
Number of participants with abnormal laboratory values and/or adverse events that are related to treatment. | Baseline up to Week 30 post first dose
Number of participants with treatment-related adverse events. | Baseline up to Week 30 post first dose
Number of participants with changes in the physical examination findings. | Baseline to Week 30 post first dose

SECONDARY OUTCOMES:
Mean change from baseline in pulmonary capillary wedge pressure (PCWP). | Baseline to Week 24 post first dose
  Measured by RHC between those who received TX000045 and those with placebo.
Mean change from baseline in PVR for all participants. | Baseline to Week 24 post first dose
  Measured by RHC between those who received TX000045 and those with placebo.
Mean change from baseline in cardiac output (CO) for all participants and in participants with CpcPH. | Baseline to Week 24 post first dose
  This is measured by RHC between those who received TX000045 and those with placebo.
Mean change from baseline in exercise capacity in all participants and in participants with CpcPH. | Baseline to Week 30 post first dose
  This is measured by mean change from baseline in 6-minute walk test (6MWT) distance between those who received TX000045 and those with placebo.
Mean change from baseline in total pulmonary resistance (TPR) for all participants and in participants with CpcPH. | Baseline to Week 24 post first dose
  This is measured by RHC between those who received TX000045 and those with placebo.
Mean change from baseline in mean pulmonary arterial pressure (mPAP) for all participants and in participants with CpcPH. | Baseline to Week 24 post first dose
  This is measured by RHC between those who received TX000045 and those with placebo.
Mean change from baseline in N-terminal pro-brain natriuretic peptide (NT-proBNP) for all participants and in participants with CpcPH between those who received TX000045 and those with placebo. | Baseline to Week 30 post first dose
Mean change from baseline responses on the Kansas City Cardiomyopathy Questionnaire (KCCQ) for all participants and in participants with CpcPH. | Baseline to Week 24 post first dose
  To evaluate the effect of TX000045 vs. Placebo on Kansas City Cardiomyopathy Questionnaire (KCCQ) scores. Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a validated tool to assess quality of life in patients with heart failure. It contains 4 subdomains: physical limitation, symptom frequency, QOL, and social limitations. Each subdomain provides an individual score from 0 to 100, with 0 denoting the worst and 100 the best possible health status.
Evaluate the incidence of immunogenicity of TX000045 by the number of participants with detectable anti-drug antibody titers. | Day 1, Week 2, Week 4, Week 8, Week 16, Week 24 and Week 30 post first dose
Number of participants with change in antibody titers following treatment with TX000045 (Immunogenicity). | Day 1, Week 2, Week 4, Week 8, Week 16, Week 24 and Week 30 post first dose

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rogers, MD, Study Director — Tectonic Therapeutic
Locations (78):
- United States (30):
  - Phoenix, Phoenix, Arizona
  - Scottsdale, Scottsdale, Arizona
  - San Francisco, San Francisco, California
  - Santa Rosa, Santa Rosa, California
  - Aurora, Aurora, Colorado
  - Jacksonville, Jacksonville, Florida
  - Tampa, Tampa, Florida
  - Augusta, Augusta, Georgia
  - McDonough, McDonough, Georgia
  - Boise, Boise, Idaho
  - Chicago, Chicago, Illinois
  - Indianapolis, Indianapolis, Indiana
  - USA, Louisville, Kentucky
  - Baltimore, Baltimore, Maryland
  - Boston, Boston, Massachusetts
  - Minneapolis, Minneapolis, Minnesota
  - St Louis, St Louis, Missouri
  - Omaha, Omaha, Nebraska
  - New York, New York, New York
  - Durham, Durham, North Carolina
  - Toledo, Toledo, Ohio
  - Philadelphia, Philadelphia, Pennsylvania
  - Pittsburgh, Pittsburgh, Pennsylvania
  - York, York, Pennsylvania
  - Rock Hill, Rock Hill, South Carolina
  - Port Arthur, Port Arthur, Texas
  - Waco, Waco, Texas
  - Salt Lake City, Salt Lake City, Utah
  - United States, Norfolk, Virginia
  - Richmond, Richmond, Virginia
- Yerevan, Yerevan, Armenia
- Australia (11):
  - Camperdown, Camperdown, New South Wales
  - Macquarie, Macquarie, New South Wales
  - New Lambton, New Lambton, New South Wales
  - Sydney, Sydney, New South Wales
  - Wollongong, Wollongong, New South Wales
  - Auchenflower, Auchenflower, Queensland
  - Chermside, Chermside, Queensland
  - Hobart, Hobart, Tasmania
  - Malvern, Malvern, Victoria
  - Camperdown, Camperdown
  - New Lambton, New Lambton
- Austria, Vienna, Austria
- Belgium (2):
  - Brussel, Brussels
  - Genk, Genk
- Bulgaria (3):
  - Pleven, Pleven
  - Plovdiv, Plovdiv
  - Sofia, Sofia
- Georgia (2):
  - Tbilisi, Tbilisi, Tb
  - Tbilisi, Tbilisi
- Mainz, Mainz, Germany
- Riga, Riga, Latvia
- Chisinau, Chisinau, Moldova
- New Zealand (2):
  - Christchurch, Christchurch
  - Dunedin, Dunedin
- Poland (6):
  - Białystok, Bialystok
  - Krakow, Krakow
  - Łodź, Lodz
  - Lublin, Lublin
  - Warsaw, Warsaw
  - Wrocław, Wroclaw
- Portugal (3):
  - Almada, Almada
  - Lisboa, Lisbon
  - Porto, Porto
- Romania (3):
  - Bucuresti, Bucharest
  - Craiova, Craiova
  - Targu Mures, Târgu Mureş
- Serbia (5):
  - Nis, Belgrade, Belgrade, Nis
  - Belgrade, Belgrade
  - Serbia, Belgrade
  - Sremska Kamenica, Kamenitz
  - Kragujevac, Kragujevac
- Spain (5):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Santiago de Compostela ( Coruña ), Santiago de Compostela
  - Toledo, Toledo
  - Valencia, Valencia
- Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No